CLINICAL TRIAL: NCT04848701
Title: Anterior Uterocervical Angle for Latent Phase Duration in Post Term Pregnancies
Brief Title: Uterocervical Angle: a Screening Tool That Estimates the Latent Phase Duration in Post Term Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecolog, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20.11.31
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Post Term Pregnancy
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- uterocervical angle (Other): uterocervical angle is the angle between lower segment of uterus and cervix
  Interventions: Other: latent phase duration; Other: uterocervical angle (UCA)

INTERVENTIONS:
Other: latent phase duration — latent phase duration in post term pregnancies
Other: uterocervical angle (UCA) — uterocervical angle is the angle between lower segment of uterus and cervix

SUMMARY:
To evaluate the performance of uterocervical angle (UCA) in the prediction of latent phase duration in post term pregnancies

ELIGIBILITY:
Inclusion Criteria:

* Patients with singleton pregnancies
* Post term pregnancies
* Patients with vertex presentation,
* Patients with intact membranes
* Patients with no uterine contractions

Exclusion Criteria:

* women with BMI >30,
* multiparity and multiple pregnancies,
* patients with macrosomia (>4500 gr),
* patients with major fetal congenital abnormality or fetal death and any contraindications to vaginal birth (e.g. active genital herpes),
* patients with abnormal Pap smears,
* patients with a history of previous cesarean section, myomectomy, hysteroscopic surgeries, dilatation and curettages, loop electrosurgical excision procedures, and cervical conization.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
prediction of latent phase duration by uterocervical angle in post term pregnancies | 5 months
  In patients diagnosed with late term pregnancy, the uterocervical angle and cervical length were measured by transvaginal ultrasound (TVUS) at the time of admission to the delivery room before labor induction.

SECONDARY OUTCOMES:
the relative success of UCA in active phase and duration of labor prediction in post term pregnancies | 5 months
  5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı Yenigül, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No